CLINICAL TRIAL: NCT02199431
Title: Interventional, Open-label, Interaction Study Investigating the Effects of Itraconazole (Inhibitor of CYP3A4/5) on the Pharmacokinetics and Safety and Tolerability of Lu AF11167 in Healthy Young Subjects
Brief Title: Study to Evaluate the Effect of a Known and Marketed Product, Itraconazole (Mycosis Treatment) on Lu AF11167 Entering the Body and Subsequently Elimination. The Study is a Drug-drug Interaction Study in Healthy Volunteers.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 14380A; 2013-003870-28 (EudraCT Number)
Record Dates: First submitted 2014-07-23; First posted 2014-07-24 (Estimated); Last update posted 2015-09-21 (Estimated); Status verified 2015-09

CONDITIONS: Healthy
Keywords: Lu AF11167; Interaction
MeSH Terms: interventions — Itraconazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lu AF1167 capsule 0.5 mg (Experimental): Single oral dose (day 1)
  Interventions: Drug: Lu AF11167
- Lu AF11167 0.5 mg capsule + itraconazole 200 mg capsule (Experimental): Itraconazole administered once daily for 7 days (day 3-9); Lu AF11167 administered as a single dose on day 8
  Interventions: Drug: Lu AF11167; Drug: Itraconazole

INTERVENTIONS:
Drug: Lu AF11167
Drug: Itraconazole
  Arms: Lu AF11167 0.5 mg capsule + itraconazole 200 mg capsule

SUMMARY:
The purpose of this study is to evaluate the increase in exposure of Lu AF11167 following a single oral dose of Lu AF11167 with and without administration of multiple oral doses of itraconazole (a strong CYP3A4/5 inhibitor) in healthy subjects with inferred metabolic status as CYP2C19 extensive metabolisers

ELIGIBILITY:
Inclusion Criteria:

* Subjects be 18 years of age and 55 years of age and with a BMI >18.5 kg/m2 and <30.0 kg/m2 at the Screening Visit. Women must not be pregnant or lactating.

Other pre-defined inclusion and exclusion criteria may apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-07; Primary Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Area under the Lu AF11167 plasma concentration-time curve from zero to infinity (AUC0-inf) | Day 1 and 8
Maximum observed plasma concentration (Cmax) of Lu AF11167 | Day 1 and 8

SECONDARY OUTCOMES:
Area under the Lu AF36201 plasma concentration-time curve from zero to infinity (AUC0-inf) | Day 1 and 8
Maximum observed plasma concentration (Cmax) of Lu AF36201 | Day 1 and 8

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- Covance, Leeds, United Kingdom